CLINICAL TRIAL: NCT01305148
Title: Warfarin Adverse Event Reduction For Adults Receiving Genetic Testing at Therapy INitiation (WARFARIN)
Acronym: WARFARIN
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor is raising funds for the remainder of the study
Sponsor: Iverson Genetic Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IG-0109
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Anti-coagulation Therapy; DVT; Pulmonary Embolism; Joint Surgery Multiple; Atrial Fibrillation; Prosthetic Replacement of Mitral Valve
Keywords: warfarin; genetic testing; personalized medicine; anti-coagulants; coumadin
MeSH Terms: conditions — Pulmonary Embolism; Atrial Fibrillation | interventions — Pharmacogenomic Testing; Precision Medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Randomized - Genetic (Experimental): Subjects who are randomized to 90 days of follow-up and whose warfarin dose was determined using the genetic information from the GenoSTAT test and clinical information through the warfarindosing.org website
  Interventions: Device: Warfarin GenoSTAT Test
- Randomized - Clinical (No Intervention): Subjects who are randomized to 90 days of follow-up and whose warfarin dose was determined using the genetic information from clinical information alone through the warfarindosing.org website
- Registry (Experimental): Subjects who are followed 30 days of follow-up and whose warfarin dose was determined using the genetic information from the GenoSTAT test and clinical information through the warfarindosing.org website
  Interventions: Device: Warfarin GenoSTAT Test

INTERVENTIONS:
Device: Warfarin GenoSTAT Test — Use of genetic information from the GenoSTAT test to determine the warfarin dose
  Other Names: Warfarin GenoSTAT; pharmacogenetic testing; personalized medicine
  Arms: Randomized - Genetic; Registry

SUMMARY:
The WARFARIN Study is a clinical trial designed to determine if the use of genetic information related to warfarin sensitivity can help create a dose of warfarin that will result in less hospitalizations and deaths related to warfarin.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 65 years old
2. Beginning warfarin (0 - 3 doses of warfarin taken at the time of enrollment) for a variety of diseases or conditions that require at least 30 days oral anticoagulation with target INR ≥ 2.0

Exclusion Criteria:

1. Unable to complete the study materials (questionnaires) with or without assistance (for example, those with dementia)
2. A previous genetically determined warfarin dose
3. The treating physician does not agree to use the recommended warfarin dose or feels that the patient should not be enrolled in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3800 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of warfarin related clinical events | 30 days
  To determine if using warfarin-related pharmacogenetic information in calculating warfarin doses will change the incidence of warfarin-related clinical events, including major hemorrhage and thromboembolic events, at 30 days after initial dose, when compared to warfarin doses calculated without pharmacogenetic data.

SECONDARY OUTCOMES:
INR Tests | 30 days
  Comparison of the number of INR tests performed before warfarin dose stabilization (i.e. two consecutive INR tests within the target range)
Warfarin Doses | 90 days
  Comparison of the cumulative warfarin dose necessary to reach warfarin dose stabilization (i.e. two consecutive INR tests within the target range)
Hemorrhagic Events | 90 days
  The number of major hemorrhagic adverse events at 60 and at 90 days separately after warfarin initiation
Minor hemorrhagic events | 90 days
  The number of minor hemorrhagic adverse events at 30, 60 and at 90 days separately after warfarin initiation
Major thromboembolic events | 90 days
  The number of major thromboembolic adverse events at 60 and at 90 days separately after warfarin initiation for
INR tests | 30 days
  The percentage of the total INR tests performed in the first 30 days which are out of target range
SF-12 | 90 days
  The overall, Physical Composite Score (PCS) and Mental Composite Score (MCS) of the SF-12 quality of life questionnaire at 30 days and at 90 days separately after warfarin initiation
Prescriber adherence | 30 days
  Prescriber adherence to dosing recommendations through subject interview and comparison of dose recommendation to dose prescribed for the first four doses of warfarin

CONTACTS AND LOCATIONS:
Overall Officials: An Pang Chieng, MD, Principal Investigator — Alhambra Hospital
Locations (56):
- United States (56):
  - Veterans' Affairs Medical Center, Birmingham, Alabama
  - Cardiovascular Consultants - Thunderbird, Glendale, Arizona
  - Cardiovascular Consultants - Phoenix, Phoenix, Arizona
  - Orthoarkansas, Little Rock, Arkansas
  - Comprehensive Cardiovascular Specialists, Alhambra, California
  - St. Joseph's Medical Center, Stockton, California
  - Colorado Heart & Vascular, Denver, Colorado
  - Okaloosa Heart & Vascular, Crestview, Florida
  - Infinity-Northshore, Fort Lauderdale, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Heart Rhythm Specialists, Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Grady Hospital, Atlanta, Georgia
  - Cardiology of Atlanta, Atlanta, Georgia
  - Atlanta Heart Group, Decatur, Georgia
  - Southern Heart Research Institute, Riverdale, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Rockford Cardiovascular Research Foundation, Rockford, Illinois
  - Carle Foundation, Urbana, Illinois
  - Community Hospital Anderson, Anderson, Indiana
  - St. Mary's, Evansville, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - NECCR, Falls River, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Thoracic and Cardiovascular Institute, Lansing, Michigan
  - Kansas City Heart Foundation, Kansas City, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Billings Clinic, Billings, Montana
  - Nebraska Heart Institute, Grand Island, Nebraska
  - Nebraska Heart, Lincoln, Nebraska
  - Alegent, Omaha, Nebraska
  - Hackensack Medical Center, Hackensack, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Mission Hospital, Asheville, North Carolina
  - Sanford Health Research, Fargo, North Dakota
  - Aultman Hospital, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Corvallis Clinic, Corvallis, Oregon
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Carolina Cardiology, Rock Hill, South Carolina
  - St. Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Nexxus Research, Bedford, Texas
  - Legacy Heart Center, Plano, Texas
  - Scott & White, Temple, Texas
  - Providence Health Network, Waco, Texas
  - Intermountain Medical Center, Murray, Utah
  - Overlake Hospital, Bellevue, Washington
  - Family Health Care of Ellensburg, Ellensburg, Washington
  - Polyclinic, Seattle, Washington
  - Swedish Hospital, Seattle, Washington
  - Franciscan Research Center, Tacoma, Washington
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin